CLINICAL TRIAL: NCT06508333
Title: Efficacy and Safety of Vitamin D Supplementation Combined With Alarm Therapy in Treating Nocturnal Enuresis: A Prospective, Randomized Controlled Trial
Brief Title: Efficacy and Safety of Vitamin D Supplementation Combined With Alarm Therapy in Treating Nocturnal Enuresis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xing Liu (Other)
Responsible Party: Sponsor-Investigator, Xing Liu, Professor, Doctor, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024424
Record Dates: First submitted 2024-07-14; First posted 2024-07-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Enuresis
MeSH Terms: conditions — Enuresis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alarm therapy (Active Comparator): These patients will receive alarm therapy for 8 weeks
  Interventions: Behavioral: alarm therapy
- Alarm therapy combined with short-term high dose exogenous vitamin D supplementation (Experimental): These patients will receive high-dose vitamin D supplementation (more than 2000IU daily) and alarm therapy for 8 weeks
  Interventions: Behavioral: alarm therapy; Drug: Vitamin D3

INTERVENTIONS:
Behavioral: alarm therapy — These patients will receive alarm therapy for 8 weeks.
Drug: Vitamin D3 — These patients will receive high-dose vitamin D supplementation (more than 2000IU daily) (combined with alarm therapy) for 8 weeks.
  Arms: Alarm therapy combined with short-term high dose exogenous vitamin D supplementation

SUMMARY:
This prospective, randomized, two-arm, parallel-design controlled clinical trial aims to determine whether high-dose vitamin D supplementation combined with alarm therapy improves outcomes in children with primary monosymptomatic nocturnal enuresis compared to alarm therapy alone.

DETAILED DESCRIPTION:
Nocturnal enuresis (NE) is characterized by recurrent involuntary urination during sleep in children aged 5 years and older, persisting for over three months with at least two episodes per week. This condition, resulting from the child's inability to awaken from sleep, exhibits a prevalence rate ranging from 4.8% to 15.2%, which notably declines with age. Moreover, NE significantly impacts the psychological well-being and overall quality of life of affected individuals. The primary treatments for NE include desmopressin acetate (DDAVP) and behavioral interventions (BI). While these modalities offer therapeutic benefits, their implementation is often prolonged and fraught with challenges, including adverse drug reactions and a high rate of symptom recurrence after treatment discontinuation. These factors complicate adherence for both patients and their families.

Patients with NE are more likely to suffer from vitamin D deficiency. This study aims to determine the effect of vitamin D supplementation as an adjunctive therapy to alarm therapy in the treatment of primary monosymptomatic nocturnal enuresis(PMNE). Eligible patients aged 5-18 years with a diagnosis of NE will be randomly assigned to receive either high-dose vitamin D supplementation combined with alarm therapy or alarm therapy alone. Serum levels of 25(OH)D will be measured at baseline. Symptom severity will be assessed at baseline and follow-up, along with other sociodemographic data. This study will provide more information on the role of vitamin D supplementation in managing PMNE.

ELIGIBILITY:
Inclusion Criteria

* Children aged 5-18 years diagnosed with PMNE-defined as intermittent urinary incontinence during sleep in a children who are never dry for more than 6 months and have no other lower urinary tract symptoms-according to the latest International Children's Continence Society guidelines, presenting at outpatient urology clinics.
* Serum vitamin D level below 30 ng/mL.
* Written informed consent obtained from each participant and their guardian.
* Adequate psychological and cognitive function, no communication barriers, and ability to accurately report symptoms and potential adverse reactions during treatment.

Exclusion Criteria

* Urological malformations or serious urological disease, such as hypospadias, cryptorchidism, posterior urethral valves, vesicoureteral reflux, neurogenic bladder, urinary tumors, urinary stones, or bladder/urethral injuries.
* Neurological disorders, including epilepsy, spinal cord injury or dysplasia, spinal embolism syndrome, multiple sclerosis, autism spectrum disorder, or attention-deficit/hyperactivity disorder.
* Endocrine diseases, such as diabetes mellitus or hyperthyroidism.
* Severe systemic disease, including significant cardiac disease, renal or hepatic insufficiency, pulmonary disease, bone deformities, gastrointestinal disorders, or inherited metabolic disorders.
* Conditions predisposing to sleep apnea, such as adenoid or tonsillar hypertrophy, deviated nasal septum, craniofacial abnormalities, or central sleep apnea.
* History of gastrointestinal or urological surgery.
* Use of anticonvulsant, antiepileptic, corticosteroid, or anti-tuberculosis medications.
* History of hypercalcemia, hyperphosphatemia, or renal rickets.
* Unexplained hematuria or urinary tract infection within the past year.
* Allergy to vitamin D formulations.
* Concurrent participation in other clinical studies.
* Unwillingness to participate or poor anticipated follow-up compliance.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in enuresis frequency | 8 week
  Change in enuresis frequency from baseline to follow-up
Response after interventions | 8 weeks
  Response rate: defined as a ≥50% reduction in the number of wet nights per week
Complete response after interventions | 8 weeks
  The rate of complete response was defined as a 100% reduction in wet nights per week.

SECONDARY OUTCOMES:
Change in quality of life score | 8 week
  The quality of life was assessed using a scale ranging from 0 to 3, where a score of 0 indicated no impact on family, social, or academic life, a score of 1 indicated occasional impact, a score of 2 indicated significant impact, and a score of 3 indicated severe impact on family, social, or academic life.
Change in vitamin D level | 8 week
  Change in vitamin D level from baseline to follow-up
Change in serum levels of calcium | 8 weeks
  Change in serum levels of calcium from baseline to follow-up
Global perception of improvement | 8 week
  Global perception of improvement (much better; better; about the same; worse)
Wish to receive another form of treatment? | 8 week
  Wish to receive another form of treatment? (YES; No)
Treatment adherence | 8 week
  The extent to which a patient adheres to their medication schedule, including both timing and dosage, or follows the prescribed treatment regimen
Incidence of side effects | 8 week
  Type and frequency of side effects during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xing Liu, Doctor, Study Director — Children's Hospital of Chongqing Medical University
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Apart from the participant's personal information.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 8 weeks
Access Criteria: Apart from the participant's personal information

REFERENCES:
- [Background] Wen JG, Wang QW, Chen Y, Wen JJ, Liu K. An epidemiological study of primary nocturnal enuresis in Chinese children and adolescents. Eur Urol. 2006 Jun;49(6):1107-13. doi: 10.1016/j.eururo.2005.11.011. Epub 2005 Dec 27. PMID 16406243
- [Background] Robson WL. Clinical practice. Evaluation and management of enuresis. N Engl J Med. 2009 Apr 2;360(14):1429-36. doi: 10.1056/NEJMcp0808009. No abstract available. PMID 19339722
- [Background] Hara T, Ohtomo Y, Endo A, Niijima S, Yasui M, Shimizu T. Evaluation of Urinary Aquaporin 2 and Plasma Copeptin as Biomarkers of Effectiveness of Desmopressin Acetate for the Treatment of Monosymptomatic Nocturnal Enuresis. J Urol. 2017 Oct;198(4):921-927. doi: 10.1016/j.juro.2017.04.088. Epub 2017 Apr 28. PMID 28457803
- [Background] Jorgensen CS, Horsdal HT, Rajagopal VM, Grove J, Als TD, Kamperis K, Nyegaard M, Walters GB, Eethvarethsson VO, Stefansson H, Nordentoft M, Hougaard DM, Werge T, Mors O, Mortensen PB, Agerbo E, Rittig S, Stefansson K, Borglum AD, Demontis D, Christensen JH. Identification of genetic loci associated with nocturnal enuresis: a genome-wide association study. Lancet Child Adolesc Health. 2021 Mar;5(3):201-209. doi: 10.1016/S2352-4642(20)30350-3. Epub 2021 Jan 15. PMID 33453761
- [Background] Tsuji S, Suruda C, Kimata T, Kino J, Yamanouchi S, Kaneko K. The Effect of Family Assistance to Wake Children with Monosymptomatic Enuresis in Alarm Therapy: A Pilot Study. J Urol. 2018 Apr;199(4):1056-1060. doi: 10.1016/j.juro.2017.11.072. Epub 2017 Nov 23. PMID 29175540
- [Background] Yeung CK, Sihoe JD, Sit FK, Diao M, Yew SY. Urodynamic findings in adults with primary nocturnal enuresis. J Urol. 2004 Jun;171(6 Pt 2):2595-8. doi: 10.1097/01.ju.0000112790.72612.0a. PMID 15118427